CLINICAL TRIAL: NCT01814852
Title: A Prospective, Randomized, Double Blind With Sham Control, Clinical Study to Assess the Safety and Efficacy of Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT) by 'Renova' in Patients With Erectile Dysfunction
Brief Title: Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT) by 'Renova' for Patients With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Initia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RENO-006B-MR
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Vasculogenic Erectile Dysfunction
Keywords: Low Intensity Shockwave; Extracorporeal shockwave therapy; Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shockwaves (Experimental): 4 weekly sessions of low-intensity shockwave therapy
  Interventions: Device: Shockwave system
- Control Group (Sham Comparator)
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Shockwave system
  Other Names: Renova
  Arms: Shockwaves
Device: Sham treatment — Sham treatment that looks, sounds and feels like real LI-ESWT treatment by Renova.
  Arms: Control Group

SUMMARY:
This is a prospective, randomized, double-blind clinical study for assessing the safety and efficacy of the treatments performed with Renova (LI-ESWT) on symptomatic ED patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind clinical study comparing safety and efficacy of the treatments performed with Renova (LI-ESWT) on symptomatic ED patients to the safety and efficacy of the control sham patients. Patients are randomized in a 1:1 ratio of Renova to the sham control group.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Vasculogenic ED for at least 6 months
* International Index of Erectile Function 6 (IIEF-EF) between 11 to 25
* Positive response to PDE5-I (able to penetrate on demand, Responders)
* Negative response to PDE5-I (unable to penetrate on demand even with maximum PDE5-I dosage,Non-responders)
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Psychogenic ED
* Neurological pathology
* Hormonal pathology
* Past radical prostatectomy
* Recovering from cancer during last 5 years
* Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Radiotherapy in pelvic region

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the IIEF-EF (International Index of Erectile Function- Erectile Function Domain) score at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment

SECONDARY OUTCOMES:
Change from baseline in the OSS (Overall Sexual Satisfaction) Questions 13 and 14 at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment
Change from baseline in the HES (Erection Hardness Score) at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Uri Gur, M.D., Principal Investigator
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Goyal NK, Garg M, Goel A. Re: Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study: Y. Vardi, B. Appel, A. Kilchevsky and I. Gruenwald. J Urol 2012; 187: 1769-1775. J Urol. 2012 Nov;188(5):2018-9. doi: 10.1016/j.juro.2012.07.052. Epub 2012 Sep 20. No abstract available. PMID 22999553
- [Background] Rosen RC, Cappelleri JC, Gendrano N 3rd. The International Index of Erectile Function (IIEF): a state-of-the-science review. Int J Impot Res. 2002 Aug;14(4):226-44. doi: 10.1038/sj.ijir.3900857. PMID 12152111
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209